CLINICAL TRIAL: NCT02321956
Title: Ultrasound Study of the Airway to Predict Endotracheal Tube Size in Anesthetized Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Raviwon Atisook, department of anesthesiology, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: RAti-001
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Pediatric General Anesthesia With Endotracheal Tube
Keywords: ASA class 1,2; age 1-6 years; General anesthesia with ETT
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed envelops were used. Ultrasonographers were masked with the group of patients. Participants were masked with the techniques of selecting endotracheal tubes. Care providers and outcome assessors were masked with the techniques of selecting. endotracheal tubes

ARMS (2):
- Ultrasound (Experimental): Using ultrasound measurement of the subglottic area to choose endotracheal tube size
  Interventions: Diagnostic Test: Ultrasound
- Formula (No Intervention): Using Cole's formula to choose endotracheal tube size

INTERVENTIONS:
Diagnostic Test: Ultrasound — Using ultrasound to determine the size of endotracheal tube
  Arms: Ultrasound

SUMMARY:
The purpose of this study is to determine whether ultrasound study of the airway to predict endotracheal tube size in anesthetized pediatric patients better than the tube size formula

DETAILED DESCRIPTION:
This study is to compare the methods of selecting uncuffed endotracheal tube size in pediatric patients between conventional age-based formula and ultrasound measurement of subglottic diameter.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-6 Years
* ASA class 1-2
* Elective Surgery
* GA with oral uncuff endotracheal tube

Exclusion Criteria:

* Potential difficult air way from history and physical exam
* Allergy ti ultrasound gel
* neck mass
* unstable vital sign

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proper size of endotracheal tube | 1 year
  Clinically fit of endotracheal tube with leak at 20-25 cmH2O

SECONDARY OUTCOMES:
Correlation of subglottic diameter and proper size endotracheal tube | 1 year
  Correlation of subglottic diameter measured by ultrasound and proper size endotracheal tube determined by clinically fit.

CONTACTS AND LOCATIONS:
Overall Officials: Raviwon Atisook, Principal Investigator — Department of anesthesiology siriraj hospital
Locations (1):
- Raviwon Atisook, Bangkok, Bangkoknoi, Thailand

REFERENCES:
- [Background] Shibasaki M, Nakajima Y, Ishii S, Shimizu F, Shime N, Sessler DI. Prediction of pediatric endotracheal tube size by ultrasonography. Anesthesiology. 2010 Oct;113(4):819-24. doi: 10.1097/ALN.0b013e3181ef6757. PMID 20808208